CLINICAL TRIAL: NCT02055131
Title: a Comparative Study of Aspirin Either at Fixed Dose or at a Dose Titrated by Platlet Function Analyzer(PFA-100) vs Placebo in Primary Prevention of Vascular Access for Hemodialysis
Brief Title: Antiaggregation in Primary Prevention of Vascular Access for Hemodialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Ben Salah Manel, nephrologist, Tunis University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 913
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Thrombosis
Keywords: vascular access; hemodialysis; aspirin resistance; PFA-100
MeSH Terms: conditions — Thrombosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aspirn fixed dose (Placebo Comparator): patients of this arm will receive 100 mg of aspirin daily.over the period of follow up we will detect all thromboembolic events.
  Interventions: Drug: aspirin
- aspirin dose titrated with PFA-100 (Placebo Comparator): patients of this arm will receive 100 mg of aspirin daily.this dose will be multiplied whenever the PFA-100 is not suitable.once the time of occlusion is correct ,we will keep the same dose of aspirin and continue monitoring the PFA-100 durin the follow up period.
  Interventions: Drug: aspirin
- placebo arm (No Intervention): in this group of patients we will just supervise thromboembolic events of the vascular access.

INTERVENTIONS:
Drug: aspirin
  Arms: aspirin dose titrated with PFA-100; aspirn fixed dose

SUMMARY:
This is a prospective study consisting in testing whether systematic use of aspirin is beneficial for primary prevention of vascular access for hemodialysis attested by doppler ultrasound exam. The investigators will study aspirin resistance in the population of patients undergoing hemodialysis. The investigators will test sensibility of resistant patients to aspirin dose escalation. PFA-100 is the biologic test used in this study to define aspirin resistance.

DETAILED DESCRIPTION:
Three groups of dialysed patients will be included in this study. The first is the placebo group, the second is the aspirin group fixed dose and the last group includes patients receiving a dose of aspirin titrated by the result of PFA-100.

At the end of this study the investigators will be able to identify whether systematic antiaggregation is suitable for a vascular access for hemodialysis. The investigators will also conclude which is better for patients fixed dose or aspirin dose escalation determined by the result of PFA-100. The study will analyse the prevalence of aspirin resistant patients in this particular population of dialysed patients.

ELIGIBILITY:
Inclusion Criteria:

* dialysed patients
* vascular access aged less than one year
* no serious complication of the vascular access previously such as hemorrhagic complication and tight stenosis

Exclusion Criteria:

* pregnant and breastfeeding women
* patients receiving at baseline other antiaggregant or anticoagulant
* patient not allowed to be treated by aspirin
* systolic blood pressure> 200 mmhg
* diastolic blood pressure>115 mmhg
* liver failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
number of fistula thrombosis in patients receiving a dose of aspirin titrated by the result of PFA-100 compared to placebo and fixed dose aspirin | 1 year
  patients undergoing hemodialysis via native fistula will receive either placebo or aspirin titrated dose by the PFA-100 or aspirin fixed dose to prevent thrombosis of the access .the follow up period will be fixed at 1 year and all thromboembolic complications of the access will be noted

SECONDARY OUTCOMES:
number of aspirin resistant patients even to aspirin escalation dose titrated by PFA-100 in the population of dialysed patients. | 1 year

OTHER OUTCOMES:
incidence and severity of aspirin complications in dialysed patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, professor, Study Director
Locations (1):
- clinical and medical investigation in emergency medecine laboratry,hospitalo-university center of Monastir, Monastir, Monastir Governorate, Tunisia